CLINICAL TRIAL: NCT00156624
Title: Local Taxan With Short Time Contact for Reduction of Restenosis in Distal Arteries (Thunder - Trial)
Brief Title: Thunder Trial - Local Taxan With Short Time Contact for Reduction of Restenosis in Distal Arteries
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Herzzentrum Bad Krotzingen (Unknown); Humboldt-Universität zu Berlin (Other); University of Greifswald (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Pac-2
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2006-04-25 (Estimated); Status verified 2005-09

CONDITIONS: Arterial Occlusive Diseases
Keywords: Intervention; Peripheral Vascular Disease; Drug; Restenosis; 18 years and above
MeSH Terms: conditions — Arterial Occlusive Diseases; Peripheral Vascular Diseases | interventions — Angioplasty, Balloon

INTERVENTIONS:
Drug: Balloon Angioplasty with or without drug administration

SUMMARY:
The Thunder Trail is a randomized , double-blinded, placebo controlled German multi-centre study on the efficacy of local paclitaxel for prevention of restenosis in the superficial and popliteal artery.

DETAILED DESCRIPTION:
Drug eluting stents have been proven to reduce the restenosis rate in the coronary arteries. Unfortunately drug eluting stents failed to demonstrate superiority over bare stents in the superficial femoral artery. We could show that a non-stent based delivery of Taxan was equal or superior to drug eluting stents in an animal model. This was both true for the coronary arteries and peripheral vessels.

In a prospective blinded trail >135 patients are randomized either to receive Taxan locally administered with a balloon catheter during balloon angioplasty, or together with contrast media. One group serves as control. There were no limitations due to lesion length. Follow-up angiography will be after 6 months, 12 months and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Chronic Occlusions and stenosis (history at least 6 weeks) ≥70 % diameter Stenosis > 2cm in the arteria femoralis superficialis or arteria poplitea
* Various criteria assuring ethical issues and follow up

Exclusion Criteria:

* Conditions requiring different treatment or raising serious safety concern regarding the procedure or the required medication.
* Pregnancy can not be excluded
* Doubts in the willingness or capability of the patient to allow 6 months follow up

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135
Dates: Start 2004-07; Study Completion 2007-10

PRIMARY OUTCOMES:
Late lumen loss of vessel segment following dilatation after 6 months

SECONDARY OUTCOMES:
Thrombotic complications or revascularization of the target vessel, death; adverse reactions known to occur after paclitaxel (high dose tumor therapy except reactions to the detergent)
Paclitaxel plasma concentration will be determined immediately after administration

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Tepe, MD, Principal Investigator — University Hospital of Tuebingen; Gunnar Tepe, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital of Tuebingen, Tübingen, Germany

REFERENCES:
- [Derived] Tepe G, Schnorr B, Albrecht T, Brechtel K, Claussen CD, Scheller B, Speck U, Zeller T. Angioplasty of femoral-popliteal arteries with drug-coated balloons: 5-year follow-up of the THUNDER trial. JACC Cardiovasc Interv. 2015 Jan;8(1 Pt A):102-8. doi: 10.1016/j.jcin.2014.07.023. PMID 25616822
- [Derived] Tepe G, Zeller T, Schnorr B, Claussen CD, Beschorner U, Brechtel K, Scheller B, Speck U. High-grade, non-flow-limiting dissections do not negatively impact long-term outcome after paclitaxel-coated balloon angioplasty: an additional analysis from the THUNDER study. J Endovasc Ther. 2013 Dec;20(6):792-800. doi: 10.1583/13-4392R.1. PMID 24325695
- [Derived] Tepe G, Zeller T, Albrecht T, Heller S, Schwarzwalder U, Beregi JP, Claussen CD, Oldenburg A, Scheller B, Speck U. Local delivery of paclitaxel to inhibit restenosis during angioplasty of the leg. N Engl J Med. 2008 Feb 14;358(7):689-99. doi: 10.1056/NEJMoa0706356. PMID 18272892